CLINICAL TRIAL: NCT00404729
Title: Phase 4 Study of Evaluation of Neural Conduction Along the Visual Pathways Before and After Oral Treatment With Citicoline in Patients With Optic Nerve Diseases
Brief Title: Neural Conduction Along the Visual Pathways After Oral Treatment With Citicoline in Patients With Optic Nerve Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Principal Investigator, Dr. Vincenzo Parisi, MD, Fondazione G.B. Bietti, IRCCS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 86216880; 85356727 (Other: FGBBIETTI)
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Glaucoma; Optic Neuropathy, Ischemic; Visual Pathway Disorder; Optic Nerve; Neural Conduction
Keywords: Glaucoma; Optic Neuropathy, Ischemic; Visual Pathways,; Optic nerve; Neural conduction
MeSH Terms: conditions — Glaucoma; Optic Neuropathy, Ischemic | interventions — Cytidine Diphosphate Choline

ARMS (1):
- Citicoline treatment (Other): Ten OAG patients will be untreated (NT-AOG, 10 eyes), while 20 OAG patients (T-AOG, 20 eyes) and 15 NION patients (T-NION, 14 eyes) were treated with Citicoline (oral treatment:1600 mg/die per 60 days)
  Interventions: Drug: Citicoline

INTERVENTIONS:
Drug: Citicoline — Ten OAG patients will be untreated (NT-AOG, 10 eyes), while 20 OAG patients (T-AOG, 20 eyes) and 15 NION patients (T-NION, 14 eyes) were treated with Citicoline (oral treatment:1600 mg/die per 60 days)

SUMMARY:
In the management of glaucoma, as for as in other optic nerve diseases, an important goal of ophthalmologists is represented by the possibility of influencing visual function.

In this regard, Parisi et al [Ophthalmology 1999; 106:1126-1134.] suggested the intramuscular treatment with Cytidine-5-diphosphocholine (CDP-Choline or citicoline) to improve glaucomatous visual defects. In particular, recent studies reported the effects of citicoline on glaucomatous retinal and postretinal visual structures evaluated by electrophysiological examinations (PERG and VEP). It was observed that a 2-month period of treatment with citicoline may induce improvement in both ganglion cell function (PERGs with increase in amplitudes and shortening in times-to-peak) and in neural conduction along postretinal visual pathways (VEPs with increase in amplitudes and shortening in times-to-peak). The effects of citicoline on glaucomatous retinal and postretinal structures were not present 8 months after the end of treatment. However, performing several 2-month period of treatment with citicoline during a total period of 8 years, it was found a additional improvement of the glaucomatous retinal and postretinal impairment [Parisi V. Doc Ophthalmol. 2005 Jan;110:91-102). In this work, the investigators aimed to assess whether there similar visual function outcomes can be reached by the oral treatment with citicoline in patients affected by glaucomatous optic nerve disease as of as in other optic nerve diseases (i.e. non-arteritic ischemic optic neuropathy)

DETAILED DESCRIPTION:
Participants: 30 patients with open-angle glaucoma (OAG) and 15 patients (mean age 64.6±3.3ys) with non-arteritic ischemic optic neuropathy (NION) were enrolled enrolled.

Ten OAG patients will be untreated (NT-AOG, 10 eyes), while 20 OAG patients (T-AOG, 20 eyes) and 15 NION patients (T-NION, 14 eyes) were treated with Citicoline (oral treatment:1600 mg/die per 60 days) (Cebrolux®, Tubilux, Italy).

Methods: In T-OAG, NT-OAG and T-NION patients, Visual Evoked Potentials (VEPs)were recorded in response to 15' checkerboard pattern stimuli.

VEPs were assessed 5 times during a total period of 360 days: at baseline conditions (0 day), after two different cycles of 60 days of treatment (days 0-60 and days 180-240), and after two different cycles of 120 days of wash out (days 60-180 and 240-360). In NT-AOG patients, VEPs were assessed at baseline conditions (0 day) and after 60, 180, 240 and 360 days.

ELIGIBILITY:
Inclusion Criteria:

Glaucoma Patients:

* IOP > 23 mmHg and < 28 mmHg (average of the two highest readings of the daily curve, from 8:00 a.m. to 6:00 p.m., six independent readings, one every two hours) without medical treatment;
* HFA with MD < - 2 dB; CPSD > +2 dB; fixation losses, false positive rate and false negative rate each less than 20%;
* best corrected visual acuity of 20/20 or better;
* one or more papillary signs on conventional color stereo-slides: the presence of a localized loss of neuroretinal rim (notch), thinning of the neuroretinal rim, generalized loss of optic rim tissue, optic disc excavation, vertical or horizontal cup/disc ratio greater than 0.5, cup-disc asymmetry between the two eyes greater than 0.2, peripapillary splinter hemorrhages;
* refractive error (when present) between -1.00 and +1.00 spherical equivalent;
* no previous history or presence of any disease involving cornea, lens, macula or retina;
* no previous history or presence of diabetes, optic neuritis, any disease involving the visual pathways;
* pupil diameter > 3 mm without mydriatic or miotic drugs.

Patients with non-arteritic ischemic optic neuropathy:

* IOP < 21 mmHg HFA with MD < - 2 dB; CPSD > +2 dB; fixation losses, false positive rate and false negative rate each less than 20%;
* refractive error (when present) between -1.00 and +1.00 spherical equivalent;
* no previous history or presence of any disease involving cornea, lens, macula or retina;
* no previous history or presence of diabetes of any further disease involving the visual pathways;
* pupil diameter > 3 mm without mydriatic or miotic drugs.

Exclusion Criteria:

All other condition that may influence Visual Evoked Potentials:

- previous history or presence of any disease involving cornea, lens, macula or retina or optic nerve (i.e inflammatory diseases)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-02-28 (Actual); Primary Completion 2006-02-28 (Actual); Study Completion 2006-07-30 (Actual)

PRIMARY OUTCOMES:
VEPs responses | 24 months
  P100 Implicit time and N75-P100 Amplitude

SECONDARY OUTCOMES:
Visual Field Defects | 24 months
  Humphrey 24/1: Mean Deviation and Corrected Pattern Standard Deviation

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Parisi, MD, Study Director — Fondazione G.B. Bietti-IRCCS, Rome, Italy
Locations (2):
- Italy (2):
  - Fondazione G.B. Bietti- IRCCS, Rome
  - Fondazione G.B. Bietti-IRCCS, Rome

REFERENCES:
- [Result] Parisi V. Electrophysiological assessment of glaucomatous visual dysfunction during treatment with cytidine-5'-diphosphocholine (citicoline): a study of 8 years of follow-up. Doc Ophthalmol. 2005 Jan;110(1):91-102. doi: 10.1007/s10633-005-7348-7. PMID 16249960
- See also: Fondazione G.B. Bietti-IRCCS activity (in italian language) — http://www.fondazionebietti.it